CLINICAL TRIAL: NCT03242967
Title: Phase 3, Randomized, Open Label, Active Controlled Study Evaluating the Efficacy and Safety of Three Times Per Week (TIW) Oral Dosing of Vadadustat for the Treatment of Anemia in Subjects With Dialysis-Dependent Chronic Kidney Disease (DD-CKD) (TRILO2GY)
Brief Title: Study to Evaluate Three Times Per Week (TIW) Oral Dosing of Vadadustat for Anemia in Subjects With Dialysis-Dependent Chronic Kidney Disease (DD-CKD)
Acronym: TRILOGY
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Revised study design.
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0023
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Anemia; Dialysis-Dependent Chronic Kidney Disease
Keywords: Anemia; hemoglobin; darbepoetin alfa; TIW; hypoxia-inducible factor prolyl-hydroxylase inhibitor; HIF-PHI; AKB-6548; vadadustat; renal; hypoxia-inducible factor; HIF; dialysis-dependent chronic kidney disease; CKD; DD-CKD; kidney; erythropoiesis stimulating agent; ESA
MeSH Terms: conditions — Anemia | interventions — vadadustat; Darbepoetin alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vadadustat (Experimental): Oral tablet
  Interventions: Drug: Vadadustat
- Darbepoetin alfa (Active Comparator): subcutaneous or intravenous
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Vadadustat — Oral tablet
  Other Names: AKB-6548
  Arms: Vadadustat
Drug: Darbepoetin alfa — subcutaneous or intravenous
  Other Names: Aranesp
  Arms: Darbepoetin alfa

SUMMARY:
This is a Phase 3 Study to Evaluate Three Times Per Week (TIW) Oral Dosing of Vadadustat for Anemia in Subjects with Dialysis-Dependent Chronic Kidney Disease (DD-CKD)

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age
* Receiving chronic maintenance in-center hemodialysis (3 times per week) for end-stage kidney disease
* Currently maintained on ESA therapy
* Mean screening Hb between 8.0 and 11.0 g/dL (inclusive)

Exclusion Criteria:

* Anemia due to a cause other than CKD or presence of active bleeding or recent blood loss
* Sickle cell disease, myelodysplastic syndromes, bone marrow fibrosis, hematologic malignancy, myeloma, hemolytic anemia, thalassemia, or pure red cell aplasia
* Red blood cell transfusion within 4 weeks prior to or during screening
* Anticipated to recover adequate kidney function to no longer require hemodialysis during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Mean change in Hb between baseline and the primary evaluation period | Baseline visit, Week 36
  Mean change in hemoglobin will be evaluated

SECONDARY OUTCOMES:
Mean change in Hb between baseline and the secondary evaluation period | Baseline visit, Week 52
  Mean change in hemoglobin will be evaluated
Proportion of subjects with mean Hb within the target range during the primary evaluation period | Baseline visit, Week 36
  Hemoglobin values within the target range will be evaluated
Adverse Events (AEs) and Serious Adverse Events (SAEs) | 52 weeks
  Adverse Events (AEs) and Serious Adverse Events (SAEs) will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (1):
- Research Site, Northridge, California, United States

IPD SHARING:
Plan to Share IPD: Undecided